CLINICAL TRIAL: NCT03724552
Title: Evaluation of LED Therapeutic Effect in Youth and Adults With Autism Spectrum Disorder: An Open-Label Pilot Study of a Novel Approach
Brief Title: Photobiomodulation in Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tolga A Ceranoglu, Associate Psychiatrist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002826
Record Dates: First submitted 2018-10-02; First posted 2018-10-30 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: photobiomodulation
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial LED Therapy (Participants ages 9-17) (Experimental): Transcranial Laser Emitting Diode (LED) Therapy (TLT) is a noninvasive intervention in which near-infrared light (830nm-850nm) is applied to forebrain.
  Interventions: Device: Transcranial LED Therapy (Participants ages 9-17)
- Transcranial LED Therapy (Participants ages 18-59) (Experimental): Transcranial Laser Emitting Diode (LED) Therapy (TLT) is a noninvasive intervention in which near-infrared light (830nm-850nm) is applied to forebrain.
  Interventions: Device: Transcranial LED Therapy (Participants ages 18-59)

INTERVENTIONS:
Device: Transcranial LED Therapy (Participants ages 9-17) — Transcranial Laser Emitting Diode (LED) Therapy (TLT) is a noninvasive intervention in which near-infrared light (830nm-850nm) is applied to forebrain.
  Arms: Transcranial LED Therapy (Participants ages 9-17)
Device: Transcranial LED Therapy (Participants ages 18-59) — Transcranial Laser Emitting Diode (LED) Therapy (TLT) is a noninvasive intervention in which near-infrared light (830nm-850nm) is applied to forebrain.
  Arms: Transcranial LED Therapy (Participants ages 18-59)

SUMMARY:
The purpose of this 8-week open-label study is to assess the tolerability, safety, and efficacy of Transcranial LED Therapy in patients with Autism Spectrum Disorder (ASD). The investigators propose to enroll up to 30 subjects of both genders ages 9-59 years with intact intellectual functions who meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for Autism Spectrum Disorder (ASD).

ELIGIBILITY:
Subjects may be included in the study only if they meet all of the following criteria:

* Male or female participants between 9 and 59 years of age (inclusive)
* Fulfills DSM-5 diagnostic criteria for autism spectrum disorder as established by the clinical diagnostic interview.
* Participants with at least moderately severity of ASD symptoms as demonstrated by SRS raw score ≥ 85 and CGI-ASD severity score ≥ 4
* Participants must understand the nature of the study. If the participant is under the age of 18, the participant's parent/guardian must sign an IRB-approved informed consent form before initiation of any study procedures. Participants ages 18-59 must sign an IRB-approved informed consent form before the initiation of any study procedures.
* Participants must have a level of understanding sufficient to communicate with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Participant experiencing a major psychiatric disorder will be allowed to participate in the study provided they do not meet any exclusionary criteria.
* Women of child-bearing potential must use a double-barrier method for birth control (e.g. condoms with spermicide) if sexually active.
* The subject is willing to participate in this study.

Subjects will be excluded from the study for any of the following reasons:

* Impaired intellectual capacity (clinically determined)
* Participant is unable to communicate due to delay in, or total lack of, spoken language development (grossly impaired language skills)
* Clinically unstable psychiatric conditions or judged to be at serious safety risk to self (suicidal risk) or others (within past 30 days).
* Subjects currently (within past 30 days) experiencing significant symptoms of major psychiatric disorders as clinically determined.
* Subjects with an unstable medical condition (that requires clinical attention).
* Active suicidal or homicidal ideation, as determined by clinical screening.
* The subject has a significant skin condition at the procedure sites (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo).
* The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised AVM, implantable shunt - Hakim valve).
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (in US: Visudine (verteporfin) - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid (ALA)- for non-melanoma skin cancer)
* Current treatment with a psychotropic medication on a dose that has not been stable for at least 4 weeks prior to initiating study treatment.
* Investigator and his/her immediate family, defined as the investigator's spouse, parent, child, grandparent, or grandchild.

Ages: 9 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tolga A Ceranoglu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceranoglu TA, Cassano P, Hoskova B, Green A, Dallenbach N, DiSalvo M, Biederman J, Joshi G. Transcranial Photobiomodulation in Adults with High-Functioning Autism Spectrum Disorder: Positive Findings from a Proof-of-Concept Study. Photobiomodul Photomed Laser Surg. 2022 Jan;40(1):4-12. doi: 10.1089/photob.2020.4986. Epub 2021 Dec 23. PMID 34941429

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcranial LED Therapy (Participants Ages 9-17) | Transcranial LED Therapy (Participants Ages 18-59)
Started | 0 | 12
Completed | 0 | 10
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Zero participants ages 9-17 enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial LED Therapy (Participants Ages 9-17) | Transcranial LED Therapy (Participants Ages 18-59) | Total
Number analyzed (Participants) | 0 | 10 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 10 | 10
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 9 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 10 | 10
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 1 | 1
  White |  | 8 | 8
  More than one race |  | 1 | 1
  Unknown or Not Reported |  | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in ASD Symptoms Social Responsiveness Scale 2 (SRS-2) Scale.
Description: Change in ASD symptoms as measured by change from baseline on the Social Responsiveness Scale 2 (SRS-2) scale.
  The SRS-2 is a 65-item rating scale completed that is used to measure the severity of autism spectrum symptoms as they occur in natural settings. The SRS-2 School Age form is completed by a parent or guardian for patients ages 9-17 and the SRS-2 Adult Self-report is completed by patients ages 18-59. Total raw scores range from 0 to 195, with higher scores indicating increased symptom severity.
Time Frame: Baseline to 8 weeks
Population: Zero participants ages 9-17 enrolled
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Transcranial LED Therapy (Participants Ages 9-17) | Transcranial LED Therapy (Participants Ages 18-59)
Number analyzed (Participants) | 0 | 10
scores on a scale |  | -30.6 (17.9)

2. Primary Outcome: Number of Participants With CGI Improvement Scores of ≤ 2 at Week 8
Description: The Clinical Global Impression Improvement scale (CGI-ASD-I) is a clinician rated measure of ASD improvement. Improvement scores range from 1 (very much improved) to 7 (very much worse).
Time Frame: 8 weeks
Population: Zero participants ages 9-17 enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Transcranial LED Therapy (Participants Ages 9-17) | Transcranial LED Therapy (Participants Ages 18-59)
Number analyzed (Participants) | 0 | 10
Participants |  | 7

ADVERSE EVENTS:
Time Frame: 8 weeks (from baseline to end of study)
Arm/Group | Transcranial LED Therapy (Participants Ages 9-17) | Transcranial LED Therapy (Participants Ages 18-59)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial LED Therapy (Participants Ages 9-17) (N=0) | Transcranial LED Therapy (Participants Ages 18-59) (N=10)
Insomnia (Nervous system disorders) | NA | 1 (2)
Headache (Nervous system disorders) | NA | 2 (5)
Warmth at Application Site (General disorders) | NA | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT03724552/Prot_SAP_000.pdf